CLINICAL TRIAL: NCT02509013
Title: Prevalence of Chronic Kidney Disease and Its Association With Clinical Outcome in Patients With Coronary Heart Disease: a Prospective, Multi-center, Hospital-based Study
Brief Title: Prevalence of Chronic Kidney Disease and Its Association With Clinical Outcome in Patients With Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Other Study IDs: WI198103
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Heart Disease; Chronic Kidney Disease
Keywords: chronic kidney disease; stable coronary heart disease; prevalence
MeSH Terms: conditions — Coronary Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, multi-center, hospital-based observational study. The aim of the study is to evaluate the prevalence of chronic kidney disease in patients with stable coronar heart disease.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the prevalence of chronic kidney disease(CKD) in patients with stable coronary heart disease. The secondary aims include: 1. To evaluate the awareness of CKD in patients with stable coronary heart disease. 2. To find out risk factors that is associated with CKD in these patients. 3. To evaluate the association between CKD and cardiovascular events during one-year's follow-up. Based on sample size estimation, the plan is to recruit 10000 patients from 100 centers. Patients who participate the study will finish one-year's follow up (0 day, 6 months and 12 months after recruitment). During the baseline visit, patients' demographic characters will be collected, and laboratory tests will be performed for urinalysis, renal function, hepatic function, etc. During the 6 months' follow up, MACE(Major adverse cardiovascular events) will be recorded through phone or face to face interview between investigators and patients. MACE include all-cause mortality, cardiovascular mortality, non-fatal myocardial infarction, documented re-hospitalization for unstable angina pectoris, and coronary revascularization (including percutaneous coronary intervention and CABG). During the 12 month's follow up, MACE will be recorded, and laboratory tests will be performed again.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years.
* Patients with clinical evidence of stable coronary heart disease, who meet at least one of the following three criterias:

  a. Stable coronary heart disease with objective evidence of atherosclerosis, either coronary angiography shows ≥50% stenosis of at least one of the coronary main stems or first-level branches, or typical exertional angina pectoris with positive stress tests(ECG stress test, echocardiograph stress test, or stress radionuclide myocardial imaging). b Diagnosed of myocardial infarction at least 3 months before recruitment. c.Coronary revascularization(PCI or CABG) at least 3 months before recruitment.
* Informed consent signed by patients or legal guardians.
* Willing to and capable of being followed up for 1 year.

Exclusion Criteria:

* Non-atherosclerotic coronary heart disease
* Deterioration of heart failure during the past 3 months
* Exposed to contrast agent during the past one month.
* History of amputation
* Pregnancy
* Female patients in menstrual period(still eligible after menstrual period)
* Organ failure other than heart failure and kidney failure
* Comorbid other diseases, and life expectancy <1 year
* Considered not fit for the study due to other reasons, including but not restricted to : a. Severe infection; b. Acute kidney injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 eligible sites over the country will participate. Each site will recruit patients who fit the inclusion standard in chronological order
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of chronic kidney disease in patients with stable coronary heart disease | 1 year
  After recruitment, urinalysis, urine albumin/creatinine ratio(ACR), and serum creatitine will be tested. Chronic kidney disease is defined as ≥1 of the following abnormalities: 1)estimated GFR<60ml/min per1.73m2. The eGFR is estimated using the CKD-EPI equation ; 2) Presence of proteinuria. Proteinuria is defined as urine ACR >30mg/g, or urinalysis showing positive proteinuria.

SECONDARY OUTCOMES:
the awareness rate of chronic kidney disease in patients with stable coronary heart disease | 1 year
factors associated with chronic kidney disease in patients with stable coronary heart disease | 1 year
  The participants will be divided into two groups based on whether CKD is present. Means and proportions will be used to describe the baseline characteristics(e.g. gender, age, history of hypertension, diabetes mellitus, dyslipidemia, and laboratory results, etc.) . T tests and chi-square tests will be used to test differences between CKD group and non-CKD group, to explore factors that are associated with the presence of CKD. Independent associations between presence of CKD and individual characteristics will be assessed using multivariable logistic models.
the association between CKD and cardiovascular events during one-year's follow-up | 2 year
  The rate of occurrence of MACE after one-year's follow-up will be described in the CKD group and non-CKD group. Univariate and multivariate cox proportional hazard model will be used to analyze whether the presence of CKD is an independent risk factor for the occurrence of MACE one year after.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No